CLINICAL TRIAL: NCT02409758
Title: The Effectiveness of the Comprehensive Voice Rehabilitation Program Compared With Vocal Function Exercises Method in Behavioral Dysphonia: A Randomized Controlled Clinical Trial.
Brief Title: Comprehensive Voice Rehabilitation Program Compared With Vocal Function Exercises
Acronym: Voicetherapy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Vanessa Pedrosa Vieira, PhD, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010/15166-3; 2010/15166-3 (Other: FAPESP - Brazil)
Record Dates: First submitted 2015-03-19; First posted 2015-04-07 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Dysphonia
Keywords: Voice disorders; Hoarseness; Therapy
MeSH Terms: conditions — Dysphonia; Voice Disorders; Hoarseness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- VFE voice therapy (Active Comparator): Voice therapy: Vocal Function Exercises applied during 6 weeks
  Interventions: Behavioral: Voice therapy
- CVRP voice therapy (Experimental): Voice therapy: Comprehensive Voice Rehabilitation Program applied during 6 weeks
  Interventions: Behavioral: Voice therapy

INTERVENTIONS:
Behavioral: Voice therapy — Voice therapy applied during 6 weeks.
  Other Names: Voice treatment; SLP

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of the Comprehensive Voice Rehabilitation Program compared with Vocal Function Exercises in behavioral dysphonia.

DETAILED DESCRIPTION:
Introduction: Voice therapy is the best indication for the most voice disorders, with a strong degree of recommendation based on systematic reviews and randomized clinical trials, with a predominance of benefit over risk. Some speech therapy techniques are specific, others are organized principles or with eclectic approaches, that use a combination of strategies. So far, few studies have tested the effectiveness of treatment for dysphonia due to time spent, safety and improved quality of life more comprehensive as they are made in clinical. Objective: To evaluate the effectiveness and safety of the Comprehensive Voice Rehabilitation Program compared with Vocal Function Exercises in behavioral dysphonia. Methods: 106 professional of voice with dysphonia behavior, between 18 and 50 years old and vocal complaints for more than six months. These professionals have been evaluated by an otolaryngologist, randomized to participate of Vocal Function Exercises arm or Comprehensive Voice Rehabilitation Program arm. Both arms were follow for six sessions with speech therapists and reassessed when finish the period and after one month. The primary outcomes assessed are: reduction of VHI score, improved voice quality in the CAPE-V and improves the larynx condition. Conclusions: The Comprehensive Voice Program has an eclectic approach and follows the philosophy of what is practiced in clinics in Brazil. We believe this program can demonstrate the power of voice therapy effectiveness more organized to solve problems, with shorter duration of treatment, benefit patient health and funding agencies such as Unified Public Health System (SUS) and health insurance.

ELIGIBILITY:
Inclusion Criteria:

* voice professionals with behavioral dysphonia, with or without larynx lesions, with otorhinolaryngologist's indication;
* over 6 months with vocal complain;
* 3 or more signs and symptoms in the questionary.

Exclusion Criteria:

* Other kind of vocal disorder, speech or language disorder, malignant lesions, hormonal disturbances related by the patient, laryngeal papilloma, etc.
* Singers;
* neurological problems;
* acute larynx problem.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Improvement of the vocal quality (assessed by two self assessment questionnaires) | First assesment in the beggining of the treatment; 2nd assesment after 6 weeks of treatment; 3rd assesment a month after the end of treatment.
  The improvement was assessed by two questionnaires of self assessment vocal quality: Voice Related Quality of life questionnaire (VRQOL) and Voice Handicap Index (VHI) in the three different moments: pre therapy, post therapy and one month after therapy

SECONDARY OUTCOMES:
Perceptual auditory analysis (assessed by 3 senior SLP) | First assesment in the beggining of the treatment; 2nd assesment after 6 weeks of treatment; 3rd assesment a month after the end of treatment.
  The general grade of hoarseness was assessed blindness by 3 senior SLP in the three different moments: pre therapy, post therapy and one month after therapy. The 3 SLP assessors was blinded according to kind of therapy and moment of evaluation.
Improvement of larynx (evaluation by blind assessor) | First assesment: in the beggining of the treatment; 2nd assesment: after 6 weeks of treatment; 3rd assesment: a month after the end of treatment.
  Evaluation of the larynx by a senior otorhinolaryngologist in the three different moments: pre therapy, post therapy and one month after therapy. The otorhinolaryngologist assessor was blinded according to the kind of therapy and moment of evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa P Vieira, PhD, Study Chair — Federal University of São Paulo

REFERENCES:
- [Background] Ziegler A, Gillespie AI, Abbott KV. Behavioral treatment of voice disorders in teachers. Folia Phoniatr Logop. 2010;62(1-2):9-23. doi: 10.1159/000239059. Epub 2010 Jan 8. PMID 20093840
- [Result] MacKenzie K, Millar A, Wilson JA, Sellars C, Deary IJ. Is voice therapy an effective treatment for dysphonia? A randomised controlled trial. BMJ. 2001 Sep 22;323(7314):658-61. doi: 10.1136/bmj.323.7314.658. PMID 11566828
- [Result] Niebudek-Bogusz E, Sznurowska-Przygocka B, Fiszer M, Kotylo P, Sinkiewicz A, Modrzewska M, Sliwinska-Kowalska M. The effectiveness of voice therapy for teachers with dysphonia. Folia Phoniatr Logop. 2008;60(3):134-41. doi: 10.1159/000120290. Epub 2008 Mar 12. PMID 18334848